CLINICAL TRIAL: NCT04835870
Title: Zanubrutinib Combination With R-CHOP in Treating Patients With Newly Diagnosed Untreated Non-GCB DLBCL
Brief Title: Zanubrutinib Plus R-CHOP for Patients With Newly Diagnosed Untreated Non-GCB DLBCL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZR-CHOP
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-03

CONDITIONS: Non-GCB/ABC Diffuse Large B-Cell Lymphoma
Keywords: Zanubrutinib, R-CHOP, Newly diagnosed Non-GCB DLBCL
MeSH Terms: interventions — zanubrutinib; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- R-CHOP + Zanubrutinib (Experimental): Zanubrutinib plus Rituximab, Cyclosphosphamide, Doxorubicin, Vincristine and Prednisone (R-CHOP)
  Interventions: Drug: Zanubrutinib; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone

INTERVENTIONS:
Drug: Zanubrutinib — Zanubrutinib-160mg bid PO d0-d20(1-21d)
  Other Names: BTK inhibitors
Drug: Rituximab — Rituximab-375 mg/m2 i.v d0 (/21d)
  Other Names: MabThera
Drug: Cyclophosphamide — Cyclophosphamide-750 mg/m2 i.v d1 (/21d)
  Other Names: CTX
Drug: Doxorubicin — Doxorubicin-50 mg/m2 i.v d1 (/21d)
  Other Names: ADM
Drug: Vincristine — Vincristine-1.4 mg/m2 i.v d1 (/21d)(2 mg max)
  Other Names: VCR
Drug: Prednisone — Prednisone-100 mg p.o d1-d5 (/21d)
  Other Names: Prednisonum

SUMMARY:
Aim of this study will evaluate the efficacy and safety of zanubrutinib in combination with R-CHOP for newly diagnosed untreated Non-GCB DLBCL Patients

DETAILED DESCRIPTION:
Diffuse large B-cell lymphoma (DLBCL) is the most common type of non-Hodgkin's lymphoma. According to Hans' algorithms, DLBCL can be identified as 2 subtypes: germinal b-cell-like(GCB) and non-germinal b-cell-like(non-GCB). Approximately 50 to 60% of DLBCL was non-GCB subtype DLBCL.The non-GCB DLBCL revealed poor clinical outcomes. Bruton's tyrosine kinase (BTK) inhibitors have established therapeutic activity in B cell malignancies, with potential activity in non-GCB DLBCL. This study will evaluate the efficacy and safety of zanubrutinib in combination with R-CHOP for newly diagnosed untreated Non-GCB DLBCL Patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed Non-GCB DLBCL with extrinsic involvement
2. Age ≥ 18 years
3. Measurable disease of at least 15mm(node)/10mm（extranodal）
4. ECOG performance status 0-2
5. Adequate organ function:Cardiac ejection fraction (EF) ≥ 50%;Creatinine clearance rate (≥30 mL/min) of serum creatinine; Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) ≤3 times ULN
6. Adequate bone marrow function:Platelet count (≥ 50×10^9/L);Hemoglobin (≥ 8 g/dL);The absolute value of neutrophils (≥1.0×10^9/L)
7. Estimated survival time ≥3 months
8. Subjects of child-bearing or child-fathering potential must be willing to practice birth control from the time of enrollment on this study until the follow-up period of the study

Exclusion Criteria:

1. Accepted major surgery within 4 weeks before treatment;
2. Diagnosis of primary mediastinal lymphoma or primary CNS lymphoma;
3. Previous history of indolent lymphoma;
4. Prior malignancy (other than DLBCL), except for cured malignant tumors with no active lesions for 3 years;Adequate treatment of inactive lesions in non-melanoma skin cancer 、malignant tonsilloma or carcinoma in situ;
5. History of intracranial haemorrhage in preceding 6 months,requires or receiving anticoagulation with warfarin or equivalent antagonists;
6. Requires treatment with a strong/medium CYP3A inducer;
7. The previous use of anthracycline-based drugs > 150 mg/m2;
8. Evidence of complications or medical conditions, including but not limited, that may interfere the conduct of the study or place the patient at serious risk:significant cardiovascular disease(class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification、myocardial infarction within 6 months of screening、uncontrolled or symptomatic arrhythmias) and/or significant lung disease;
9. HIV infection and/or active hepatitis B or active hepatitis C;
10. Uncontrolled systemic infection;
11. Pregnant or breasting-feeding women;
12. According to the researchers' judgment, patients' underlying condition may increase their risk of receiving research drug treatment, or confuse their judgment on toxic reactions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival(PFS) | up to 18 months
  To measure the duration of response to ZR-CHOP over a follow-up period of 18 months

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | up to 18 months
  To measure the duration of response to ZR-CHOP over a follow-up period of 18 months
Complete Response Rate | up to 18 months
  Number of patients who achieved complete response after treatment by ZR-CHOP
Duration of Response | up to 18 months
  Duration of overall response will be assessed from the first ZR-CHOP given to progression,death or last follow-up.
Overall Survival | up to 18 months
  OS will be assessed from the first ZR-CHOP given to death or last follow-up.
Adverse events profile | Measured from start of treatment until 28 days after last dose
  Number of participants with adverse events. Frequencies of toxicities based on the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 5.0 will be tabulated

CONTACTS AND LOCATIONS:
Overall Officials: Depei Wu, M.D, Study Chair — The First Affiliated Hospital of Soochow University
Locations (16):
- China (16):
  - The First Affiliated Hospital of USTC Anhui Provincial Hospital, Hefei, Anhui
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Changshu No.1 People's Hospital, Suzhou, Jiangsu
  - Suzhou Hongci Hematology Hospital, Suzhou, Jiangsu
  - Zhangjiagang First Peoples Hospital, Suzhou, Jiangsu
  - Affiliated Hospital Of Jiangnan University, Wuxi, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Shandong Provincial Hospital Affiliated to Shandong First Medical University, Jinan, Shandong

REFERENCES:
- [Derived] Geng H, Jia S, Zhang Y, Li J, Yang Q, Zeng L, Zong X, Lu Y, Lu S, Zhou J, Li C, Wu D. Efficacy and safety of zanubrutinib plus R-CHOP in treatment of non-GCB DLBCL with extranodal involvement. Front Immunol. 2023 Aug 21;14:1219167. doi: 10.3389/fimmu.2023.1219167. eCollection 2023. PMID 37671152